CLINICAL TRIAL: NCT00346580
Title: The Effects of HIV Protease Inhibitors in Severe Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1254-03
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir

SUMMARY:
Sepsis is the leading cause of death in critically ill patients in the United States. It develops in approximately 750,000 Americans annually, and more than 210,000 of them die. Despite improvements in supportive treatment, mortality has changed very little, and until recently, no sepsis-specific treatments were available. Protease inhibitors have seemed to have an immune benefit that extends beyond their ability to prevent HIV replication. T cells in those patients treated with protease inhibitors have reduced rates of death than in those patients not receiving therapy.

DETAILED DESCRIPTION:
Our hypothesis is that protease inhibitor therapy will prevent apoptosis associated with sepsis, and this will be manifested as improved clinical outcome, as assessed by 28-day mortality, APACHE II and III, and SOFA scores. All patients enrolled in the study will receive the standard of care for sepsis at Mayo Clinic Rochester. Patients will receive 1250 mg of Nelfinavir/placebo twice each day for seven days with regularly scheduled blood draws (Days 0, 4, and 7).

ELIGIBILITY:
Infection criteria:known or suspected infection, as evidenced by one or more of the following: WBC in normally sterile body fluid, radiographic evidence of pneumonia, a syndrome associated with a high risk of infection.

Modified SIRS criteria: must meet three or more of the following four criteria: a temperature higher than 38C or lower than 36C, heart rate of more than 90 beats/minute, respiratory rate of more than 20 breaths/minute (or on a mechanical ventilator), WBC more than 12,000/mm(3) or less than 4,000/mm(3).

Dysfunctional organs criteria:must meet one or more of the following five criteria:cardiovascular system dysfunction, kidney dysfunction, respiratory dysfunction, hematological dysfunction, unexplained metabolic acidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Death from any cause at 28 days and 3 months
Daily APACHE II and III scores
Daily SOFA scores

SECONDARY OUTCOMES:
Change in CD4 and CD8 T-cell apoptosis, as determined by flow cytomerty, at the time of enrollment, on Day 4 of therapy, and upon completion of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Badley, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States